CLINICAL TRIAL: NCT00067028
Title: A Prospective Randomized Phase I/II Study of Clofarabine (Clo) and Ara-C vs Clo and Ida vs Clo Plus Ida and Ara-C in Patients With First Relapse or First Salvage of Primary Refractory AML; and High-Grade MDS(>/= 10% Blasts); or CML in Myeloid Blasts Phase as Front Line Therapy or in First Salvage.
Brief Title: Clofarabine Combinations in Relapsed/Refractory Acute Myeloid Leukemia (AML), Myelodysplastic Syndromes (MDS) and Myeloid Blast Phase Chronic Myeloid Leukemia (CML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0181
Record Dates: First submitted 2003-08-08; First posted 2003-08-13 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; CML Myeloid Blast Phase; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Clofarabine; Clofarex; Clolar; Ara-C; Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Idarubicin; Idamycin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Clofarabine; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clofarabine + Ara-C (Experimental): Clofarabine 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Ara-C Starting dose: 1 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
  Interventions: Drug: Clofarabine 40mg/m^2; Drug: Ara-C 1 g/m^2
- Clofarabine + Idarubicin (Experimental): Clofarabine 22.5 mg/m^2 by vein over 1 hour daily for 5 days.
  Idarubicin 10 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Interventions: Drug: Idarubicin 10mg/m^2; Drug: Clofarabine 22.5mg/m^2
- Clofarabine + Idarubicin + Ara-C (Experimental): Clofarabine 22.5 mg/m^2 by vein over 1 hour daily for 5 days.
  Idarubicin 6 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Ara-C Starting dose: 0.75 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
  Interventions: Drug: Ara-C 0.75 g/m^2; Drug: Clofarabine 22.5mg/m^2; Drug: Idarubicin 6 mg/m^2

INTERVENTIONS:
Drug: Clofarabine 40mg/m^2 — 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Other Names: Clofarex; Clolar
  Arms: Clofarabine + Ara-C
Drug: Idarubicin 10mg/m^2 — 10 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Clofarabine + Idarubicin plus Ara-C:
  6 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Other Names: Idamycin®,; Idamycin PFS®
  Arms: Clofarabine + Idarubicin
Drug: Ara-C 0.75 g/m^2 — 0.75 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
  Other Names: Cytosar-U®; Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
  Arms: Clofarabine + Idarubicin + Ara-C
Drug: Clofarabine 22.5mg/m^2 — 22.5 mg/m^2 by vein over 1 hour daily for 5 days.
  Other Names: Clofarex; Clolar
  Arms: Clofarabine + Idarubicin; Clofarabine + Idarubicin + Ara-C
Drug: Ara-C 1 g/m^2 — 1 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
  Other Names: Cytosar-U®; Cytarabine; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
  Arms: Clofarabine + Ara-C
Drug: Idarubicin 6 mg/m^2 — 6 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Other Names: Idamycin®,; Idamycin PFS®
  Arms: Clofarabine + Idarubicin + Ara-C

SUMMARY:
The goal is to compare the drug combinations clofarabine/idarubicin/ara-C, clofarabine/ara-C, and clofarabine/idarubicin in the treatment of patients with Acute Myeloid Leukemia, high-grade MDS, or myeloid blast phase of Chronic Myeloid Leukemia who have relapsed following their initial therapy.

DETAILED DESCRIPTION:
Clofarabine is a new drug that was designed to help treat leukemia. Ara-C and idarubicin are drugs that are commonly used to help treat leukemia.

Before treatment starts, you will be asked questions about your medical history and have a complete physical exam. You will have blood samples (about 1 tablespoon) collected for routine lab tests. You will either have an echocardiogram or a multiple-gated acquisition (MUGA) scan to check on the function of your heart. You will have a sample of bone marrow collected to check on the status of the disease. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

After each cycle of therapy, you will not receive the next cycle of chemotherapy until your blood counts have recovered and any possible side effects have gone away (for around 3 to 6 weeks). If the disease gets worse or side effects become too severe, treatment will stop. You must stay in Houston for the first 4 to 6 weeks (average) of treatment and are required to return to Houston to receive each additional cycle of chemotherapy (up to 6 days each cycle).

You will be assigned to receive treatment with clofarabine plus idarubicin and ara-C.

For participants in the clofarabine/idarubicin/ara-C group, the clofarabine will be given by vein over 1 hour once a day for 5 days in a row, on Days 2 to 6 of each cycle. Idarubicin will be given by vein over 30 minutes for 3 days in a row, on Days 1 to 3 of each cycle. Ara-C will be given by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle. Idarubicin is usually started around 1 hour after the completion of clofarabine, and ara-C about 4 hours after the start of the clofarabine infusion. This 6 day period is called a cycle of chemotherapy.

You will receive at least 1 cycle of therapy. If after 1 or 2 cycles of therapy it is found that the disease is responding to therapy, you may continue to receive therapy for up to 4 additional courses of "consolidation therapy". During the "consolidation therapy" you will also be given treatment courses with ara-C alone. When ara-C is given alone it will be given as a continuous infusion, 24 hours a day, for 5 days in a row. You will be given a portable pump so that this treatment can be done as an outpatient. The combination drug courses and the ara-C courses will alternate (ara-C alone, combination, ara-C alone, combination) for a total of 4 courses. If it is found that the disease is not responding to chemotherapy, you will be taken off the study and your doctor will discuss other treatment options with you.

Before you receive each dose of drug(s), you will have a complete physical exam. During treatment, you will have blood (about 1 tablespoon) collected at least once a week during the first 2 courses of therapy, then every 2-4 weeks after. Bone marrow samples will be collected every other week during treatment to check on the status of the disease. The blood and bone marrow samples may be collected more often if your doctor feels it is necessary.

If, at any time, the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

After your last course of treatment, you will have a follow-up visit scheduled. At this visit, you will have blood (about 1 tablespoon) collected for routine tests. You will have a sample of bone marrow collected to check on the status of the disease. You will also have a repeat echocardiogram or MUGA scan to check on the function of your heart.

This is an investigational study. Clofarabine has been authorized by the FDA to be used in research only. Idarubicin and ara-C are both FDA approved and are commercially available. Up to 120 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years and < 60 years.
2. Must be in first relapse of AML, or must receive treatment as first salvage in primary refractory AML; or have high-risk MDS (>/= 10% blasts) with not more than one prior regimen of chemotherapy (therapy with hematopoietic growth factors, biological or targeted therapies are not counted). Patients in CML myeloid blast phase may receive clofarabine as frontline therapy or in first salvage.
3. Total bilirubin </= 2mg/dL, Serum glutamic pyruvic transaminase (SGPT) </= 4 upper limit of normal (ULN), creatinine </= 2.0mg/dL.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
5. Signed informed consent.
6. Male and female patients who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 7 days of study enrollment (applies only if patient is of childbearing potential. Non-childbearing is defined as >= 1 year postmenopausal or surgically sterilized).

Exclusion Criteria:

1. Previous treatment with clofarabine.
2. Active, uncontrolled, systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment, or any severe, concurrent disease, which, in the judgment of the investigator and after discussion with the Principal Investigator, would make the patient inappropriate for study entry.
3. Symptomatic central nervous system (CNS) involvement.
4. Patients who receive other chemotherapy. Patients must have been off previous therapy of >/= 2 weeks and must have recovered from acute toxicity of all previous therapy prior to enrollment. Treatment may start earlier following discussion with the Principal Investigator.
5. Cardiac ejection fraction </= 30%.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2003-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan H Faderl, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 2003 to October 2009. All participants were recruited at the University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Clofarabine + Ara-C: Clofarabine 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Ara-C :1 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
Period: Overall Study
Arm/Group | Clofarabine + Ara-C | Clofarabine + Idarubicin | Clofarabine + Idarubicin + Ara-C
Started | 17 | 36 | 63
Completed | 17 | 36 | 63
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clofarabine + Ara-C: Clofarabine 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Ara-C : 1 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
- Total: Total of all reporting groups
Arm/Group | Clofarabine + Ara-C | Clofarabine + Idarubicin | Clofarabine + Idarubicin + Ara-C | Total
Number analyzed (Participants) | 17 | 36 | 63 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 28 | 58 | 100
  >=65 years | 3 | 8 | 5 | 16
Age, Continuous [Median (Full Range); unit: years] | 55 [39 to 73] | 57 [25 to 73] | 51 [18 to 80] | 54 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 26 | 30 | 63
  Male | 10 | 10 | 33 | 53
Region of Enrollment [Number; unit: participants]
  United States | 17 | 36 | 63 | 116

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Response assessed by blood test or bone marrow aspirate following day 21 of induction and then every 2 weeks thereafter until remission or non-response. Complete remission (CR): Disappearance all clinical and/or radiologic evidence of disease; Neutrophil count > 1.0 x10^9/L and platelet count >100x10^9/L, and normal bone marrow differential (< 5% blasts). Complete remission without platelet recovery (CRp): Peripheral blood and bone marrow results as for CR, but with platelet counts of > 20 x 10^9/L and < 100 x 10^9/L. Partial remission (PR): Peripheral blood count recovery as for CR, but with decrease in marrow blasts of > 50% and not more than 6-25% abnormal cells in the marrow. All other responses considered as failures.
Time Frame: Up to 6 years
Population: Two participants in the Clofarabine + Idarubicin (CI) arm were not evaluable for response.
Measure: Number; unit: participants
Groups:
- Clofarabine + Idarubicin: Clofarabine 30 - 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Idarubicin 10 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
- Clofarabine + Idarubicin + Ara-C: Clofarabine 30 - 40 mg/m^2 by vein over 1 hour daily for 5 days.
  Idarubicin 6 mg/m^2 by vein over 30 minutes, around one hour after clofarabine, for the first 3 days of 5 day cycle.
  Ara-C Starting dose: 0.75 g/m^2 by vein over 2 hours for 5 days in a row, on Days 1 to 5 of each cycle.
Arm/Group | Clofarabine + Ara-C | Clofarabine + Idarubicin | Clofarabine + Idarubicin + Ara-C
Number analyzed (Participants) | 17 | 34 | 63
participants
  CR | 4 | 9 | 16
  CRp | 2 | 5 | 7
  PR | 0 | 1 | 1

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of participants with complete response following treatment out of all participants in that particular treatment group. Response assessed by blood test or bone marrow aspirate following day 21 of induction and then every 2 weeks thereafter until remission or non-response. Complete remission (CR): Disappearance all clinical and/or radiologic evidence of disease; Neutrophil count > 1.0 x10^9/L and platelet count >100x10^9/L, and normal bone marrow differential (< 5% blasts). Complete remission without platelet recovery (CRp): Peripheral blood and bone marrow results as for CR, but with platelet counts of > 20 x 10^9/L and < 100 x 10^9/L. Partial remission (PR): Peripheral blood count recovery as for CR, but with decrease in marrow blasts of > 50% and not more than 6-25% abnormal cells in the marrow. All other responses considered as failures.
Time Frame: Up to 6 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Clofarabine + Ara-C | Clofarabine + Idarubicin | Clofarabine + Idarubicin + Ara-C
Number analyzed (Participants) | 17 | 34 | 63
Percentage of Participants | 36 | 44 | 24

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Clofarabine + Ara-C | Clofarabine + Idarubicin | Clofarabine + Idarubicin + Ara-C
All-Cause Mortality (participants affected / at risk) | 4/17 | 3/36 | 8/63
Serious Adverse Events (participants affected / at risk) | 4/17 | 13/36 | 13/63
Other Adverse Events (participants affected / at risk) | 17/17 | 36/36 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Ara-C (N=17) | Clofarabine + Idarubicin (N=36) | Clofarabine + Idarubicin + Ara-C (N=63)
Supraventricular Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cholevystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fungal Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Infection (orbit) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection (Skin Abcess) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Prolonged Myelosuppression (General disorders) | 0 (0) | 5 (5) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Ara-C (N=17) | Clofarabine + Idarubicin (N=36) | Clofarabine + Idarubicin + Ara-C (N=63)
Nausea/Vomiting (Gastrointestinal disorders) | 17 (47) | 36 (69) | 63 (78)
Diarrhea (Gastrointestinal disorders) | 17 (47) | 36 (50) | 63 (66)
Constipation (Gastrointestinal disorders) | 17 (17) | 28 (28) | 13 (13)
Mucositis (Gastrointestinal disorders) | 17 (24) | 30 (30) | 27 (27)
Anorexia/Dyspepsia (Gastrointestinal disorders) | 17 (17) | 17 (17) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 17 (59) | 36 (63) | 39 (39)
CNS (General disorders) | 17 (24) | 36 (36) | 25 (25)
Cardiac (Cardiac disorders) | 6 (6) | 13 (13) | 10 (10)
Hepatic (Hepatobiliary disorders) | 17 (77) | 36 (52) | 63 (68)
Renal (Renal and urinary disorders) | 12 (12) | 8 (8) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes